CLINICAL TRIAL: NCT04308083
Title: The Influence of a New Implant Neck Configuration on Hard and Soft Tissue Healing. A Randomized Controlled Clinical Trial
Brief Title: The Influence of a New Implant Neck Configuration on Hard and Soft Tissue Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PerioCentrum Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sweden&Martina Prama project
Record Dates: First submitted 2019-10-27; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Implant Geometry, Osseointegration, Soft Tissue Volume, Marginal Bone Levels, Soft Tissue Recession, Volumetric Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- convergent neck (Active Comparator): Group A Sweden & Martina Prama (P). Transgingival tapering machined collar, 2.8 mm in height.
  Interventions: Procedure: dental implant placement
- divergent neck (Sham Comparator): Group B Straumann Tissue Level (TL). Transgingival widening polished collar, 1.8 mm in height.
  Interventions: Procedure: dental implant placement

INTERVENTIONS:
Procedure: dental implant placement — Implants will be placed according to the manufacturer recommendations. Implants will be placed at 1.5 to 2.0 mm from the adjacent natural tooth. However, these distances will be directed by the prosthetic crown needed and they will be recorded in the CRF.

SUMMARY:
Title: Randomized Controlled Clinical Trial comparing two dental implants with different neck configurations.

Objective: To evaluate the changes in peri-implant soft tissues and marginal bone level when using a one-piece implant with a widening transgingival machined collar and a one-piece implant with a tapering transgingival machined collar.

Design: The study will be a prospective parallel randomized clinical trial with a 12 month follow up conducted in 5 private dental practices. A total of 50 patients meeting the inclusion criteria will be randomized in one of the two groups to receive 1 single implant placed in healed ridges. Radiographic and clinical measurements will be taken post-insertion, baseline (post-loading) 6 and 12 months after loading.

Study Hypothesis: The hypothesis of this study is that there will be no differences in the preservation of the peri-implant marginal bone level and peri-implant soft tissues between the two implant neck designs.

DETAILED DESCRIPTION:
The study will be a prospective parallel randomized clinical trial (RCT) of approximately 20 months of duration, in which each patient will receive 1 implants placed in the posterior mandible. If the patients fulfill the inclusion criteria after implant site preparation, they will be randomized to either receive an implant with a one-piece tapering neck configuration (P) or with a widening neck configuration (TL).

52 patients, male or female, aged 18 or older, who are missing one tooth in the posterior mandible (positions 4-6).

A randomization list will determine which implant type has to be inserted. This randomization list will be generated by an independent investigator.

Patients will be recruited by the investigator consecutively. Prior to implant site preparation, the clinician will determine if the patient still meets the inclusion criteria at surgery in particular if the bone quantity is sufficient. Patients who do not meet the inclusion criteria will be excluded from the study and will therefore not be randomized. The patients will be randomized to receive P implant or TL implant.

For both groups, impression will be taken 8 weeks post insertion. Details with regard to the prosthetic procedures and materials used for the restoration of the implants will be provided in a separate section of this protocol.

Standardized peri-apical radiographs will be taken before and after prosthesis placement to document the crestal bone level at the day of loading.

Standardized photographs will be taken to measure the soft tissue at the time of loading.

The thickness of the soft tissue will be measured 2 mm apical to the gingival margin with a needle.

Routine controls are due at 6 and 12 months post loading. Peri-apical radiographs will be taken after implant placement, before/after loading and at 12 months post loading. Final impressions will be taken at 12 months post loading to evaluate volumetric changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old
* Each patient will have one missing tooth in the posterior mandible (positions 4-6). There must be a natural tooth mesially and distally to the implant site. Free end situation are not allowed.
* Adequate bone quality and quantity at the implant site to permit the insertion of a SWEDEN AND MARTINA® Prama Implant in the diameter of 4.25 mm and in the length of 8.5 mm, 10 mm or a Straumann Tissue Level in the diameter of 4.1 mm and in the length of 8 mm or 10mm.
* Opposing dentition must be natural teeth or teeth/implant supported fixed restoration(s).
* Patient has been informed of the follow-up visits and is willing to return to the clinical center for these follow-up visit.

Exclusion Criteria:

* These exclusion criteria might be systemic or local. In addition to the general contra-indication for dental implants the following exclusion criteria will be observed:

Systemic exclusion criteria:

* Medical conditions requiring prolonged use of steroids and/or with medications that can interfere with bone metabolism
* History of leukocyte dysfunction and deficiencies
* History of neoplasic disease requiring the use of radiation or chemotherapy
* Patients with history of renal failure
* Patients with metabolic bone disorders such as osteoporosis
* History of uncontrolled endocrine disorders
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Use of any investigational drug or device within the 30 day period immediately prior to implant surgery on study day 0
* Alcoholism or drug abuse
* History of immunodeficiency syndromes
* Patients who smoke >20 cigarettes per day or cigar equivalents.
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, unreliability

Local exclusion criteria:

* Any bone augmentation on the implant site which was performed in the previous 3 months
* Local inflammation, including untreated periodontitis
* Mucosal diseases such as erosive lichen planus
* History of local irradiation therapy
* Presence of osseous lesions
* Unhealed extraction sites (less than 6 weeks post extraction of teeth in intended sites)
* Severe bruxing or clenching habits
* Persistent intraoral infection

Exclusion criteria at surgery:

* Lack of primary stability of implant.
* Presence of vertical dehiscence
* Unable to place the implant according to the prosthetic requirements. In any of these instances the patient will not be included in the study and a new patient will be recruited and randomized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-11-17 (Estimated); Study Completion 2021-03-17 (Estimated)

PRIMARY OUTCOMES:
soft tissue volumetric changes | 1 year
  soft tissue volumetric changes between baseline and one year

SECONDARY OUTCOMES:
marginal bone levels | 1 year
  marginal bone levels between baseline and at one year
implant survival rate | 1 year
  no mobility at crown placement and at one year
probing pocket depth | 1 year
  probing pocket depth at crown placement and at one year
recession | 1 year
  recession at crown placement and at one year
keratinized mucosa | 1 year
  keratinized mucosa at crown placement and at one year

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Vignoletti, PhD, Principal Investigator — PerioCentrum Research
Locations (1):
- PerioCentrum Madrid, Madrid, Spain